CLINICAL TRIAL: NCT06735274
Title: Transcranial Doppler (TCD) Ultrasound for Predicting and Understanding Cognitive Decline in Cerebral Vascular Disease.
Brief Title: Transcranial Doppler (TCD) Ultrasound and Cognition in Cerebral Vascular Disease. (SUNRISE)
Acronym: SUNRISE
Status: Completed | Type: Observational
Sponsor: Universidade do Porto (Other)
Collaborators: Hospital de Sao Joao, Porto (Unknown); RISE Study Group (Network)
Responsible Party: Sponsor
Other Study IDs: SUNRISE
Record Dates: First submitted 2024-08-08; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Vascular Accident (CVA)/Stroke
Keywords: Ischemic Stroke; Haemorrhagic Stroke; Cerebral Vascular Disease
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke | interventions — Neurovascular Coupling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — This is a prospective cohort study with inclusion of consecutive ischemic stroke patients. The assessment conducted on the included patients will consist of a cerebral transcranial Doppler evaluation, a cognitive screening, and questions regarding functional recovery and daily living activities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Ischemic Stroke (Carotid Circulation): Patients with ischemic stroke of atherosclerotic, cardioembolic and embolic etiology from an unknown source
  Interventions: Diagnostic Test: Cerebral Autoregulation (CAR); Diagnostic Test: Neurovascular coupling (NVC); Diagnostic Test: Microembolic signals (MES); Diagnostic Test: Montreal Cognitive Assessment (MoCA); Diagnostic Test: Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE); Diagnostic Test: Instrumental Activities of Daily Living Scale (IADL); Diagnostic Test: Modified Rankin Scale for Neurologic Disability (mRS)
- Ischemic Stroke (Posterior Circulation): Patients with ischemic stroke of atherosclerotic, cardioembolic and embolic etiology from an unknown source
  Interventions: Diagnostic Test: Cerebral Autoregulation (CAR); Diagnostic Test: Neurovascular coupling (NVC); Diagnostic Test: Microembolic signals (MES); Diagnostic Test: Montreal Cognitive Assessment (MoCA); Diagnostic Test: Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE); Diagnostic Test: Instrumental Activities of Daily Living Scale (IADL); Diagnostic Test: Modified Rankin Scale for Neurologic Disability (mRS)
- Haemorrhagic Stroke: Patients with intracerebral haemorrhages
  Interventions: Diagnostic Test: Cerebral Autoregulation (CAR); Diagnostic Test: Neurovascular coupling (NVC); Diagnostic Test: Microembolic signals (MES); Diagnostic Test: Montreal Cognitive Assessment (MoCA); Diagnostic Test: Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE); Diagnostic Test: Instrumental Activities of Daily Living Scale (IADL); Diagnostic Test: Modified Rankin Scale for Neurologic Disability (mRS)

INTERVENTIONS:
Diagnostic Test: Cerebral Autoregulation (CAR) — Cerebral Autoregulation (CAR) is the mechanism capable of maintaining cerebral blood flow constant despite fluctuations in blood pressure. The evaluation of dynamic CAR (dCAR) with spontaneous blood pressure variations allows it to be applied in acute and non-collaborating patients
Diagnostic Test: Neurovascular coupling (NVC) — Neurovascular coupling (NVC) is the relationship between neural activity and cerebral blood flow, allowing this activity to be evaluated in spatiotemporal terms .
Diagnostic Test: Microembolic signals (MES) — Microembolic signals (MES)
Diagnostic Test: Montreal Cognitive Assessment (MoCA) — Montreal Cognitive Assessment (MoCA)
Diagnostic Test: Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) — Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE)
Diagnostic Test: Instrumental Activities of Daily Living Scale (IADL) — Instrumental Activities of Daily Living Scale (IADL)
Diagnostic Test: Modified Rankin Scale for Neurologic Disability (mRS) — Modified Rankin Scale for Neurologic Disability (mRS)

SUMMARY:
This study aims to contribute to the identification of factors that may be predictive of cognitive function and to provide data on cerebral hemodynamic in ischemic and haemorrhagic stroke. This study will prospectively study cerebral autoregulation, neurovascular coupling and microembolic signs in cerebrovascular patients with ischemic and haemorrhagic stroke and its relationship with cognitive function and functional recovery

ELIGIBILITY:
Inclusion Criteria:

* Minimum age limit: 18 years
* Patients with intracerebral haemorrhages; Patients with ischemic stroke of atherosclerotic, cardioembolic and embolic etiology from an unknown source;
* Previous mRS equal or more than 4;
* National Institutes of Health Stroke Scale (NIHSS)≤20 at admission;
* IQCODE final score<3.0

Exclusion Criteria:

* History of dementia or other central nervous system disease associated with cognitive impairment;
* Absence of adequate temporal bone window for Transcranial Doppler monitoring;
* Patients with a large cerebral infarct (greater than on third of the middle cerebral artery territory) or a strategic infarct (paramedian thalamus, medial frontal cortex, or hippocampus) evaluated in the 24 hours-CT;
* Average life expectancy less than 1 year for a different cause of cardiovascular disease;
* Patients with intracranial vascular malformation, intracranial venous thrombosis, head trauma or tumour and haemorrhagic transformation within an infarct;
* Serious kidney and systemic diseases;
* Active cancer patients;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes participants who suffered a stroke admitted in the stroke unit (Centro Hospitalar Universitário de São João, Porto, Portugal), being included in order of admission. Provide signed and dated informed consent; more than 18 years; Patients with intracerebral haemorrhages; Patients with ischemic stroke of atherosclerotic, cardioembolic and embolic etiology from an unknown source.
Sampling Method: Non-Probability Sample
Enrollment: 517 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Functional status | 3±1 months after onset; 12±1 months after onset
  The modified Rankin Scale (mRS):
  0 - None;
  1- No significant disability despite symptoms: able to carry out all usual duties and activities; 2 - Slight disability: unable to carry out all previous activities, but able to look after own affairs without assistance; 3 - Moderate disability: requiring some help, but able to walk without assistance; 4 - Moderately severe disability: unable to walk without assistance, unable to attend to needs without assistance; 5 - Severe disability: bed-ridden, incontinent, and requiring constant nursing care and attention; 6 - Dead
Cognitive status | 12±1 months after onset
  Cognitive status at 12 months of follow-up will be calculated based in 7-scale cognitive score operationalized from Montreal Cognitive Assessment (MoCA) together with modified Rankin Scale (mRS):
  1. - Sub-category Normal: No evidence of cognitive impairment;
  2. - Sub-category Minor Single: Scores are reduced by more than 1 point in only one cognitive domain of MoCA test;
  3. - Sub-category Minor Multi: Scores are reduced by more than 1 point in more than one cognitive domain of MoCA test;
  4. - Sub-category Major Mild: Cognitive impairments (MoCA test 20-25) and minimal functional problems (mRS less than 3);
  5. - Sub-category Major Moderate: More severe cognitive impairments (MoCA test 14-19) and more limiting function (mRS=3 or 4);
  6. - Sub-category Major Severe: Severest cognitive impairments (MoCA less than 14) and most limited function or Moderately severe/severe disability (mRS more than 4);
  7. - Sub-category Death.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Castro, PhD, Principal Investigator — Universidade do Porto
Locations (1):
- Centro Hospitalar e Universitário de São João, EPE, Porto, Portugal